CLINICAL TRIAL: NCT02252354
Title: An Open-Label, Single-Centre,Two Part Phase I Mass Balance Study to Assess the Absorption, Distribution, Metabolism, Excretion and Absolute Bioavailability of Orally Administered [14C]-TAK-385 in Healthy Male Subjects
Brief Title: TAK-385 Phase I Absorption, Distribution, Metabolism, Excretion and Absolute Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-385-1009; 2014-001564-35 (EudraCT Number); U1111-1159-5663 (Registry Identifier: WHO); 14/WA/1087 (Registry Identifier: NRES)
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — relugolix; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: [14C]-TAK-385 (Experimental): [14C]-TAK-385 80 mg, solution, orally, once on Day 1.
  Interventions: Drug: [14C]-TAK-385 Oral Solution
- Part 2: TAK-385 + [14C]-TAK-385 IV (Experimental): TAK-385 80 mg, tablets, orally, and [14C]-TAK-385 80 μg, infusion, intravenous once on Day 1.
  Interventions: Drug: TAK-385 Tablets; Drug: [14C]-TAK-385 Solution for Intravenous Infusion

INTERVENTIONS:
Drug: [14C]-TAK-385 Oral Solution — TAK-385 oral radiolabelled solution
  Arms: Part 1: [14C]-TAK-385
Drug: TAK-385 Tablets — TAK-385 tablets 2 X 40 mg
  Arms: Part 2: TAK-385 + [14C]-TAK-385 IV
Drug: [14C]-TAK-385 Solution for Intravenous Infusion — TAK-385 intravenous (IV) radiolabelled solution
  Arms: Part 2: TAK-385 + [14C]-TAK-385 IV

SUMMARY:
The purpose of this 2 part study is to look at how TAK-385 is taken up, broken down and removed from the body when given as a radiolabelled oral solution (by mouth) or as an oral tablet (by mouth) followed by a radiolabelled intravenous (IV) infusion (into the arm vein).

DETAILED DESCRIPTION:
The study will consist of 2 parts involving up to 12 healthy male participants. In Part 1, up to 6 participants will receive a single 80 mg dose of [14C]-TAK-385 administered as an oral solution. In Part 2, up to 6 participants will receive a single oral 80 mg dose of TAK-385 administered as two 40 mg tablets and an 80 μg intravenous (into a vein) dose of [14C]-TAK-385 (containing not more than 37.0kBq [1000 nCi] 14C).

This single centre study will take place in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Signs a written, informed consent form prior to the initiation of any study procedures.
2. Is a healthy male, aged 18 to 55; inclusive on Day-1.
3. Is capable of understanding and complying with protocol requirements.
4. Weighs at least 50 kg and has a body mass index (BMI) between 18.0 and 35.0 kg/m^2, inclusive at Screening or Day-1.
5. In the opinion of the investigator, is in good healthy condition on the basis of a pre-study physical examination, medical history, vital signs, electrocardiogram, and the results of blood biochemistry, hematology, and serology test and urinalysis at Screening and Day -1.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose.

Exclusion Criteria:

1. Has received any investigational compound within 45 days prior to Day -1.
2. Has received TAK-385 in a previous clinical study.
3. Has a resting systolic blood pressure ≤90 mmHg or ≥140 mmHg and a resting diastolic blood pressure ≤50 mmHg or ≥90 mmHg in supine position at Screening or Day-1.
4. QTc (Fridericia's correction) is >450 msec at Screening or at Day -1 as read on the printout of the ECG produced by the electrocardiogram (ECG) equipment and evaluated by the investigator
5. Has active liver disease or jaundice, or with alanine aminotransferase (ALT),aspartate aminotransferase (AST), or bilirubin (total bilirubin) >1.5 times the upper limit of normal (ULN) in the clinical laboratory tests at VISIT 1 and 2. The participant has positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) or known history of human immunodeficiency virus (HIV) at Screening.
6. Has a resting pulse and heart rate (as read on ECG) <45 beats per minute (bpm) or >100 bpm at Screening or Day -1.
7. Has had an acute, clinically significant illness within 30 days prior to Day -1.
8. Has a history or clinical manifestations of significant metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), hematologic, pulmonary, cardiovascular,gastrointestinal, neurological, rheumatologic, skin and subcutaneous tissue disorders,infectious, hepatic, renal, urologic, immunologic, psychiatric or mood disorders (including any past history of suicide attempt), or history of lactose intolerance.
9. Has a family history of bleeding disorders.
10. Has current or recent (within 6 months) history of gastrointestinal disease that would be expected to influence the absorption of drugs (ie, history of malabsorption,esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent heartburn, or any surgical intervention).
11. Has irregular defecation patterns (less than one defecation per two days or excessive diarrhea) and/or has a history of changes in bowel habits with daily routine or environment changes.
12. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
13. Has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic or nonperipheral vascular surgery within 6 months prior to Day - 1.
14. Has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to Day 1.
15. Has significant cardiovascular disease including, but not limited to, a history of myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, clinically significant abnormal ECGs, New York Heart Association (NYHA) Functional Classification III or IV, or documented cerebrovascular accident within 6 months prior to Day -1.
16. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 1 year prior to the Screening Visit.
17. Has used any tobacco (ie, nicotine) products (including but not limited to cigarettes, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) within 6 months prior to Day -1 or is unwilling to abstain from these products for the duration of the study or has a positive carbon monoxide test result at Screening or Day -1.
18. Has taken any medications, supplements or food products as described in the Excluded Medications section. A subject has a positive carbon monoxide test result on Day-1.
19. Has poor peripheral venous access.
20. Is unwilling or unable to comply with the protocol or scheduled appointments
21. Is unable to understand verbal and/or written English.
22. Is a study site employee, or is an immediate family member (ie, spouse, parent, child, and sibling) of a study site employee, involved in conduct of this study.
23. Has received or donated more than 400 mL of blood or blood products within the 45 days preceding the beginning of the study or plans to donate blood during the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United Kingdom from 29 September 2014 to 27 October 2014.
Pre-assignment Details: Healthy cohort of male participants were enrolled in this 2 part study, in 1 of 2 treatment groups as follows : Part 1: [14C]-TAK-385 80 milligram (mg); Part 2:TAK-385 80 mg + [14C]-TAK-385 80 microgram (mcg)
Groups:
- Part 1: [14C]-TAK-385: [14C]-TAK-385 80 mg, solution, orally, single dose on Day 1.
- Part 2: TAK-385 + [14C]-TAK-385: TAK-385 80 mg, tablets, orally, and [14C]-TAK-385 80 mcg, infusion, intravenous single dose on Day 1.
Period: Overall Study
Arm/Group | Part 1: [14C]-TAK-385 | Part 2: TAK-385 + [14C]-TAK-385
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Part 2: TAK-385 + [14C]-TAK-385 IV: TAK-385 80 mg, tablets, orally, and [14C]-TAK-385 80 mcg, infusion, intravenous single dose on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part 1: [14C]-TAK-385 | Part 2: TAK-385 + [14C]-TAK-385 IV | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Number; unit: Participants]
  Greater than(>)17 to less than equal to(<=)64 | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 5 | 6 | 11
  More than one race | 1 | 0 | 1
Caffeine Consumption [Number; unit: Participants]
  Yes | 5 | 5 | 10
  No | 1 | 1 | 2
Xanthine Consumption [Number; unit: Participants]
  Yes | 2 | 1 | 3
  No | 4 | 5 | 9
Smoking Classification [Number; unit: Participants]
  Never smoked | 5 | 3 | 8
  Current smoker | 0 | 0 | 0
  Ex-smoker | 1 | 3 | 4
Alcohol Classification [Number; unit: Participants]
  The participant has never drunk | 1 | 0 | 1
  The participant is a current drinker | 5 | 6 | 11
  The participant is an ex-drinker | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Time to Reach the Maximum Plasma and Whole Blood Radioactivity Concentration (Cmax) for [14C]-TAK-385
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax. Radioactivity corresponds to no more than (NMT) 4.7 millibecquerel (MBq) (127 microcurie [mCi]). Cmax was calculated as disintegration per minute per mL (DPM/mL). Total [14C]-TAK-385 determination of plasma and whole blood samples was determined by accelerator mass spectrometry (AMS) method.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
hours
  Whole Blood Radioactivity | 2.0 (1.4354) [0.2 to 4.0]
  Plasma Radioactivity | 2.0 (1.4354) [0.2 to 4.0]

2. Primary Outcome: Part 1: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-385
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax. Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product ([14C]-TAK-385).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
hours | 1.2 (1.4748) [0.2 to 4.0]

3. Primary Outcome: Part 1: Cmax: Maximum Observed Plasma and Whole Blood Radioactivity Concentration for [14C]-TAK-385
Description: Maximum observed concentration (Cmax) is the peak concentration of a drug after administration, obtained directly from the concentration-time curve. Radioactivity corresponds to NMT 4.7 MBq (127 mCi). Cmax was measured in nanogram equivalent per milliliter (ng eq/mL) and was calculated as disintegration per minute per mL (DPM/mL). Total [14C]-TAK-385 determination of plasma and whole blood samples was determined by AMS method.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq/mL
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
ng eq/mL
  Whole Blood Radioactivity | 45.6 (24.2)
  Plasma Radioactivity | 56.1 (34.2)

4. Primary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for TAK-385
Description: Maximum observed concentration (Cmax) is the peak concentration of a drug after administration, obtained directly from the concentration-time curve. Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product ([14C]-TAK-385).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL) | 44.7 (29.0)

5. Primary Outcome: Part 1: AUC(0-inf): Area Under the Plasma and Whole Blood Radioactivity Concentration-time Curve From Time 0 to Infinity for [14C]-TAK-385
Description: AUC(0-inf) is measure of area under the curve from time 0 to infinity. Radioactivity corresponds to NMT 4.7 MBq (127 mCi). AUC(0-inf) was measured in nanogram equivalent*hour per milliliter (ng eq*hr/mL) and was calculated as disintegration per minute per mL (DPM/mL). Total [14C]-TAK-385 determination of plasma and whole blood samples was determined by AMS method.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq*hr/mL
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
ng eq*hr/mL
  Whole Blood Radioactivity | 1521.5 (421.2)
  Plasma Radioactivity | 1771.4 (476.5)

6. Primary Outcome: Part 1: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-385
Description: AUC(0-inf) is area under the concentration-time curve from time 0 to infinity. Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product ([14C]-TAK-385) .
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
nanogram hour per milliliter (ng*hr/mL) | 382.2 (128.2)

7. Primary Outcome: Part 1: AUC(0-168): Area Under the Plasma and Whole Blood Radioactivity Concentration-Time Curve From Time 0 to 168 Hours Postdose for [14C]-TAK-385
Description: AUC(0-168) is measure of area under the curve over the dosing interval (tau),where tau is the length of the dosing interval: 168 hours in this study (AUC(0-168]). Radioactivity corresponds to NMT 4.7 MBq (127 mCi). It was calculated as disintegration per minute per mL (DPM/mL). Total [14C]-TAK-385 determination of plasma and whole blood samples was determined by AMS method.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq*hr/mL
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
ng eq*hr/mL
  Whole Blood Radioactivity | 756.5 (229.5)
  Plasma Radioactivity | 982.7 (288.7)

8. Primary Outcome: Part 1: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for TAK-385
Description: AUC(0-168) is measure of area under the curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval -168 hours in this study). Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product ([14C]-TAK-385).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
ng*hr/mL | 357.5 (119.0)

9. Primary Outcome: Part 1: Terminal Phase Elimination Half-Life (t1/2z) in Plasma and Whole Blood Radioactivity for [14C]-TAK-385
Description: Terminal phase elimination half-life (t1/2z) is the time required for half of the drug to be eliminated from the blood. Radioactivity corresponds to NMT 4.7 MBq (127 mCi). It was calculated as disintegration per minute per mL (DPM/mL). Total [14C]-TAK-385 determination of plasma and whole blood samples was determined by AMS method.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
hours
  Whole Blood Radioactivity | 285.3 (32.9) [255.9 to 333.7]
  Plasma Radioactivity | 226.1 (22.0) [192.4 to 246.1]

10. Primary Outcome: Part 1: Terminal Phase Elimination Half-Life (t1/2z) in Plasma for TAK-385
Description: Terminal phase elimination half-life (t1/2z) is the time required for half of the drug to be eliminated from the blood. Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product ([14C]-TAK-385).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
hours | 60.7 (6.6) [53.6 to 69.3]

11. Primary Outcome: Part 1: Overall Cumulative Percent Recovery of Total Dosed Radioactivity in Urine and Feces
Description: Overall cumulative percent of radioactive dose recovered in urine and feces is the total radioactivity excreted in urine and feces divided by the amount of total radioactivity dosed for each participant. Total [14-C] determination of urine and feces samples were determined by Liquid Scintillation Counting (LSC).
Time Frame: Day 1 pre-dose and various time-points (up to Day 288) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percent recovery of radioactivity
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percent recovery of radioactivity
  Urine | 4.3 (0.7)
  Feces | 82.7 (6.3)

12. Primary Outcome: Part 2: Tmax : Time to Reach the Maximum Plasma Radioactivity Concentration (Cmax) for [14C]-TAK-385
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax. Radioactivity corresponds to NMT 37.0 kilobecquerel (kBq) (1000 nanocurie [nCi]). Total radioactivity and [14C]-TAK-385 determination of plasma samples was determined by AMS.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
hours | 0.2 (0.0455) [0.1 to 0.2]

13. Primary Outcome: Part 2: Tmax : Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-385
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
hours | 2.2 (2.0897) [0.5 to 6.0]

14. Primary Outcome: Part 2: Cmax: Maximum Observed Plasma Radioactivity Concentration for [14C]-TAK-385
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Radioactivity corresponds to NMT 37.0 kBq (1000 nCi).Total radioactivity and [14C]-TAK-385 determination of plasma samples was determined by AMS.
Time Frame: Day 1 pre-dose and various time-points (up to 168hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng eq/mL | 2.6 (0.3)

15. Primary Outcome: Part 2: Cmax: Maximum Observed Plasma Radioactivity Concentration for TAK-385
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng/mL | 24.6 (13.2)

16. Primary Outcome: Part 2: AUC(0-inf): Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Infinity for [14C]-TAK-385
Description: AUC(0-inf) is measure of area under the curve from time 0 to Infinity. Radioactivity corresponds to NMT 37.0 kBq (1000 nCi).AUC(0-inf) was corrected according to Hamilton Pool result.Total radioactivity and [14C]-TAK-385 determination of plasma samples was determined by AMS.
Time Frame: Day 1 pre-dose and various sampling time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq*hr/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng eq*hr/mL | 4.2 (0.6)

17. Primary Outcome: Part 2: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-385
Description: AUC(0-inf) is measure of area under the curve from time 0 to Infinity.
Time Frame: Day 1 pre-dose and various time-points (up to 288 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng*hr/mL | 225.2 (110.8)

18. Primary Outcome: Part 2: AUC(0-168): Area Under the Plasma Radioactivity Concentration-Time Curve From Time 0 to 168 Hours Postdose for [14C]-TAK-385
Description: AUC(0-168) is measure of area under the curve over the dosing interval (tau), where tau is the length of the dosing interval :168 hours in this study (AUC(0-tau]). AUC(0-168) was corrected according to Hamilton Pool result.Radioactivity corresponds to NMT 37.0 kBq (1000 nCi).Total radioactivity and [14C]-TAK-385 determination of plasma samples was determined by AMS.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng eq*hr/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng eq*hr/mL | 3.2 (0.3)

19. Primary Outcome: Part 2: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for TAK-385
Description: AUC(0-168) is measure of area under the curve over the dosing interval (tau),where tau is the length of the dosing interval: 168 hours in this study (AUC(0-tau]). AUC was corrected using the Hamilton Pool Data to get an AUC for TAK-385.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
ng*hr/mL | 214.5 (106.3)

20. Primary Outcome: Part 2: Terminal Phase Elimination Half-Life (t1/2z) in Plasma Radioactivity for [14C]-TAK-385
Description: Terminal phase elimination half-life (t1/2z) is the time required for half of the drug to be eliminated from the blood. Radioactivity corresponds to NMT 37.0 kBq (1000 nCi).Total radioactivity and [14C]-TAK-385 determination of plasma samples was determined by AMS.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
hours | 110.5 (16.2) [96.0 to 134.5]

21. Primary Outcome: Part 2: Terminal Phase Elimination Half-Life (t1/2z) in Plasma for TAK-385
Description: Terminal phase elimination half-life (t1/2z) is the time required for half of the drug to be eliminated from the blood.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
hours | 50.6 (6.0) [42.5 to 60.3]

22. Primary Outcome: Part 2: Absolute Bioavailability for the Oral Tablet Formulation
Description: Absolute bioavailability, defined as the fraction or percentage of the unchanged, orally administered dose that is systemically available, relative to the total dose administered intravenously. AUC was corrected using the Hamilton Pool Data to get an AUC for TAK-385
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percentage bioavailability
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
percentage bioavailability | 11.6 (7.2)

23. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/F) for TAK-385
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided by AUC expressed in liters/hour (L/hr). CL which was calculated by correcting the [14C]TAK-385 AUC, following the intravenous dose with the hamilton pool result to get a true CL (L/h). Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
L/hr | 218.2 (66.7)

24. Secondary Outcome: Part 2: Apparent Oral Clearance (CL/F) for TAK-385
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided by AUC expressed in liters/hour (L/hr).CL which was calculated by correcting the [14C]TAK-385 AUC, following the intravenous dose with the hamilton pool result to get a true CL (L/h).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
L/hr | 382.9 (154.7)

25. Secondary Outcome: Part 1: Volume of Distribution (Vz/F) for TAK-385
Description: Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by the terminal elimination rate constant (λz). Plasma concentrations of TAK-385 were measured by high-performance liquid chromatography with tandem mass spectrometry method (LC-MS/MS). Correction of the LC-MS/MS derived concentrations were based upon the specific activity of the administered radiolabelled drug product.
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
Liter (L) | 18878.7 (5114.4)

26. Secondary Outcome: Part 2: Volume of Distribution (Vz/F) for TAK-385
Description: Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by the terminal elimination rate constant (λz).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
L | 28245.1 (13011.8)

27. Secondary Outcome: Part 2: Overall Cumulative Percent Recovery of Total Dosed Radioactivity in Urine and Feces
Description: Overall cumulative percent of radioactive dose recovered in urine and feces is the total radioactivity excreted in urine and feces divided by the amount of total radioactivity dosed for each participant.
Time Frame: Day 1 pre-dose and various time-points (up to 72 hours) post-dose for urine; Day 1 pre-dose and various time-points (up to 48 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percent recovery of radioactivity
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
percent recovery of radioactivity
  Urine | 13.3 (3.0)
  Feces | 22.2 (13.3)

28. Primary Outcome: Part 1: Excretion of TAK-385 and Its Metabolites in Human Feces as Percent Radioactivity
Description: Amount of total [14]C, TAK-385, metabolite A, B, and C, and others excreted from feces, calculated as percentage of recovered radioactivity, are reported. Others were calculated by subtraction of the sum of the values for TAK-385, Metabolite-A, Metabolite-B, and Metabolite-C from the value of the total radioactivity (total [14]C).Radioactivity corresponds to NMT 4.7 MBq (127 mCi).
Time Frame: 0 to 191 hours post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percentage of recovered radioactivity
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of recovered radioactivity
  Total 14[C] | 100 (0.0)
  TAK-385 | 5.1 (3.2)
  Metabolite-A | 0.3 (0.4)
  Metabolite-B | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-C | 50.6 (7.5)
  Others | 44.0 (8.1)

29. Primary Outcome: Part 1: Excretion of TAK-385 and Its Metabolites in Human Urine as Percent Radioactivity
Description: Amount of total [14]C, TAK-385, metabolite A, B, and C, and others excreted from urine, calculated as percentage of recovered radioactivity, are reported. Others were calculated by subtraction of the sum of the values for TAK-385, Metabolite-A, Metabolite-B, and Metabolite-C from the value of the total radioactivity (total [14]C).Radioactivity corresponds to NMT 4.7 MBq (127 mCi).
Time Frame: 0 to 144 hours post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percentage of recovered radioactivity
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of recovered radioactivity
  Total 14[C] | 100 (0.0)
  TAK-385 | 52.6 (19.0)
  Metabolite-A | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-B | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-C | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Others | 47.4 (19.0)

30. Primary Outcome: Part 1: Excretion of TAK-385 and Its Metabolites in Human Feces as Percentage of Dose
Description: Amount of total [14]C, TAK-385, metabolite A, B, and C, and others excreted from feces, calculated as percentage of dose. Others were calculated by subtraction of the sum of the values for TAK-385, Metabolite-A, Metabolite-B, and Metabolite-C from the value of the total [14]C.
Time Frame: 0 to 191 hours post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Total 14[C] | 80.6 (5.7)
  TAK-385 | 4.2 (2.9)
  Metabolite-A | 0.3 (0.3)
  Metabolite-B | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-C | 40.6 (4.9)
  Others | 35.6 (7.3)

31. Primary Outcome: Part 1: Excretion of TAK-385 and Its Metabolites in Human Urine as Percentage of Dose
Description: Amount of total [14]C, TAK-385, metabolite A, B, and C, and others excreted from urine, calculated as percentage of dose. Others were calculated by subtraction of the sum of the values for TAK-385, Metabolite-A, Metabolite-B, and Metabolite-C from the value of the total [14]C.
Time Frame: 0 to 144 hours post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Total 14[C] | 4.1 (0.7)
  TAK-385 | 2.2 (0.9)
  Metabolite-A | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-B | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Metabolite-C | NA (NA) — Data were not reported because none of the values were above lower limit of detection.
  Others | 2.0 (0.9)

32. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 1 Post-dose
Description: Percentage of [14]C as measured from TAK-385, metabolite A and B, and metabolite C in the plasma pools were calculated as the percentage of dose administered.
Time Frame: Hour 1 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 3 (0.7)
  Metabolite-C | 1.5 (NA)
  TAK-385 | 55.3 (0.9)

33. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 2 Post-dose
Description: as for outcome 32
Time Frame: Hour 2 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 2.5 (0.7)
  Metabolite-C | 1.2 (NA)
  TAK-385 | 68.2 (0.9)

34. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 4 Post-dose
Description: as for outcome 32
Time Frame: Hour 4 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 2.2 (0.7)
  Metabolite-C | 0.8 (NA)
  TAK-385 | 58.8 (0.9)

35. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 8 Post-dose
Description: as for outcome 32
Time Frame: Hour 8 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 3.2 (0.7)
  Metabolite-C | 1.2 (NA)
  TAK-385 | 41.5 (0.9)

36. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 12 Post-dose
Description: as for outcome 32
Time Frame: Hour 12 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 3.8 (0.7)
  Metabolite-C | 1.3 (NA)
  TAK-385 | 45.7 (0.9)

37. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 24 Post-dose
Description: as for outcome 32
Time Frame: Hour 24 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 2.6 (0.7)
  Metabolite-C | 2.1 (NA)
  TAK-385 | 53 (0.9)

38. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 36 Post-dose
Description: as for outcome 32
Time Frame: Hour 36 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 2.2 (0.7)
  Metabolite-C | 2.7 (NA)
  TAK-385 | 52.4 (0.9)

39. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 48 Post-dose
Description: as for outcome 32
Time Frame: Hour 48 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 3.2 (0.7)
  Metabolite-C | 4.5 (NA)
  TAK-385 | 48 (0.9)

40. Primary Outcome: Part 1: [14]C Distribution Profile From TAK-385 and Metabolites A, B, and C in Plasma Pools at Hour 72 Post-dose
Description: as for outcome 32
Time Frame: Hour 72 post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Number; unit: percentage of dose
Arm/Group | Part 1: [14C]-TAK-385
Number analyzed (Participants) | 6
percentage of dose
  Metabolite A and B | 3.0 (0.7)
  Metabolite-C | 3.2 (NA)
  TAK-385 | 45.9 (0.9)

41. Secondary Outcome: Part 2: Clearance (CL) for [14C]-TAK-385
Description: CL is clearance of the drug from the plasma, calculated as the drug dose divided by AUC expressed in L/hr. CL is a quantitative measure of the rate at which a drug substance is removed from the body. Radioactivity corresponds to NMT 37.0 kBq (1000 nCi).
Time Frame: Day 1 pre-dose and various time-points (up to 168 hours) post-dose
Population: PK set included all participants in the safety set with at least one measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2: TAK-385 + [14C]-TAK-385 IV
Number analyzed (Participants) | 6
L/hr | 29.4 (4.5)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (+/- 2) after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: [14C]-TAK-385 | Part 2: TAK-385 + [14C]-TAK-385 IV
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: [14C]-TAK-385 (N=6) | Part 2: TAK-385 + [14C]-TAK-385 IV (N=6)
Flatulence (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.